CLINICAL TRIAL: NCT05828459
Title: A First-in-human, Dose-escalation Followed by Expansion Study to Assess the Safety and Preliminary Efficacy of a Bispecific Antibody OT-A201 as Monotherapy and in Combination Therapy in Patients With Selected Hematological Malignancies and Solid Tumors
Brief Title: First-in-human Study of OT-A201 in Patients With Selected Hematological Malignancies and Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Onward Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A20101
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hematological Malignancy; Solid Tumor
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Immunomodulating Agents; Lenalidomide; pomalidomide; Bevacizumab; Paclitaxel; triazabicyclodecene

STUDY DESIGN:
Intervention Model Description: Monotherapy dose escalation followed by dose confirmation of combination regimens.
  Further expansion of each groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- OT-A201 monotherapy (Experimental): OT-A201 administered by IV infusion on a weekly (qw) basis. An alternative dosing schedule of every 2 weeks (q2w) may be implemented based on the clinical safety and laboratory data.
  Interventions: Drug: OT-A201
- OT-A201 in combination with iMiD (Experimental): OT-A201 in combination with lenalidomide or pomalidomide at the approved dose
  Interventions: Drug: OT-A201; Drug: IMids
- OT-A201 in combination with a specific agent (Experimental): OT-A201 in combination with late stage approved treatment (combination to be defined by a protocol amendment)
  Interventions: Drug: OT-A201; Drug: TBD Compound
- OT-A201 in combination with bevacizumab (Experimental): OT-A201 in combination with bevacizumab at the approved dose
  Interventions: Drug: OT-A201; Drug: Bevacizumab
- OT-A201 in combination with paclitaxel (Experimental): OT-A201 in combination with paclitaxel at the approved dose
  Interventions: Drug: OT-A201; Drug: Paclitaxel

INTERVENTIONS:
Drug: OT-A201 — OT-A201 IV infusion qw or q2w
Drug: IMids — Combination regimen for hematological malignancy Lenalidomide: 25 mg on Days 1 to 21 of each 28-day cycle; or Pomalidomide: 4 mg on Days 1 to 21 of each 28-day cycle
  Other Names: lenalidomide; pomalidomide
  Arms: OT-A201 in combination with iMiD
Drug: Bevacizumab — Combination regimen for solid tumor Bevacizumab: 10 mg/m² q2w
  Arms: OT-A201 in combination with bevacizumab
Drug: Paclitaxel — Combination regimen for solid tumor Paclitaxel: 175 mg/m² q3w
  Arms: OT-A201 in combination with paclitaxel
Drug: TBD Compound — Combination regimen for hematological malignancy
  Arms: OT-A201 in combination with a specific agent

SUMMARY:
This phase 1 study is aimed at establishing the safety basis of OT-A201 in the treatment of hematological malignancies and solid tumors. In the dose of escalation part it is to characterize the overall safety and tolerability profile and determine the recommended dose(s) of OT-A201 as monotherapy, and in various combination regimens. Preliminary information about anti-cancer activity will be further explored in the expansion part of the study.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically or cytologically confirmed relapsed/refractory hematological malignancy or advanced/metastatic solid cancer
* Measurable disease
* Have had all available therapeutic standards for their disease
* Willingness to undergo baseline biopsy/bone marrow aspiration in case biopsy was not collected after completion of the most recent prior therapy
* ECOG performance status ≤ 1
* Life expectancy > 3 months as assessed by the investigator
* Acceptable clinical lab results

Main Exclusion Criteria:

* Systemic steroids at a daily dose of > 10 mg of prednisone or equivalent within 28 days before study treatment. Transient use of steroids for other medical condition may be allowed
* Ongoing immune-related adverse events irAEs and or AEs ≥ grade 2 from previous therapies not resolved except vitiligo, stable neuropathy up to grade 2, hair loss, and stable endocrinopathies with substitutive hormone therapy
* Within 4 weeks of major surgery
* Documented history of active autoimmune disorder requiring systemic immunosuppressive therapy within the last 12 months
* Prior solid organ transplant
* Primary or secondary immune deficiency
* Active and uncontrolled infection requiring intravenous antibiotic or antiviral treatment
* Seropositive (except after vaccination or confirmed cure for hepatitis) for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Clinically significant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose(s) (MTD) and recommended dose(s) of OT-A201 | 28 days
  Evaluate dose-limiting toxicity (DLT) during the DLT observation period
Safety profile of OT-A201 | 6 months
  Incidence, severity, and relationship of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), TEAEs leading to discontinuation of study treatment; and clinically significant findings on clinical laboratory tests, vital signs, ECGs, and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Eric Raymond, MD, PhD, Principal Investigator — Saint-Joseph Hospital - Paris
Locations (4):
- France (4):
  - ICM - Montpellier, Montpellier
  - Saint-Eloi Hospital - Montpellier (CHU), Montpellier
  - Saint-Joseph Hospital - Paris, Paris
  - Centre Eugène Marquis, Rennes

IPD SHARING:
Plan to Share IPD: No